CLINICAL TRIAL: NCT02983955
Title: UPNRIDE Powered Wheelchair for Individuals With Walking Impairment: Evaluation of Safety and Usability
Acronym: UPNRIDE_SAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UPnRIDE Robotics Ltd. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UPNRIDE-UR-SF-01
Record Dates: First submitted 2016-11-22; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Spinal Cord Injury Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCI with Tetraplegia (Other)
  Interventions: Device: UPnRIDE Powered Wheelchair

INTERVENTIONS:
Device: UPnRIDE Powered Wheelchair — The UPnRIDE Powered Wheelchair device is a product which changes people position from sitting to standing and standing to sitting. The product provides indoor and outdoor mobility.

SUMMARY:
The UPnRIDE Powered Wheelchair device is a product which changes people position from sitting to standing and standing to sitting. The product provides indoor and outdoor mobility.

The main purpose of this study is to evaluate the safety of the UPnRIDE powered wheelchair as an outdoor and indoor mobility device by individuals with walking impairment.

DETAILED DESCRIPTION:
A new powered wheelchair has recently been developed to address the ability of the user to be able to position them in an upright, standing position. This new device is called the UPnRIDE powered wheelchair and is different from other upright wheelchairs because current standing wheelchair models have limited mobility in the standing position. The UPnRIDE is an upright or seated mobility device that is intended to provide full upright standing posture in a mobile powered wheelchair. The UPnRIDE powered wheelchair provides wheelchair and scooter users the ability to engage in society in either a standing (upright mobility) or seated position (seated mobility). Additionally, the option to have upright posture throughout the day may have the potential to improve some of the secondary medical conditions associated with the extreme sedentary lifestyle that paralysis from SCI imposes. This wheeled, motorized device can provide mobility to most urban environment situations by being able to be navigated indoors and outdoors and over different surfaces in both the standing or seated positions.

ELIGIBILITY:
Inclusion Criteria

1. Males and non-pregnant, non-lactating females
2. Ages 18-70
3. Suffered from a SCI which caused Tetraplegia, ASIA A-B-C
4. At least 1 year after SCI
5. Height of 155 to 190 cm;
6. Weight less than 100 kg
7. Able to sign informed consent.
8. Power or manual wheelchair user as a primary means of mobility
9. Regular user of a standing frame or tilt table for at least 30 minutes a week Exclusion Criteria

1. History of severe neurological disorder other than SCI (multiple sclerosis, cerebral palsy, amyotrophic lateral sclerosis, traumatic brain injury, stroke, etc.) 2. Concurrent severe medical disease 3. Pressure sores 4. Unstable spine 5. Unhealed limb or pelvic fractures 6. Psychiatric or cognitive status that may interfere with the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 3 months

SECONDARY OUTCOMES:
Successes rate of task performance | Through study completion, an average of 3 months
  Study success is defined if 70% of study subjects are defined success

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, MD, Principal Investigator — Department of Neurological Rehabilitation The Chaim Sheba Medical Center, Tel Hashomer and Sackler Faculty of Medicine,
Locations (1):
- The Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No